CLINICAL TRIAL: NCT03717337
Title: Evaluation of Success Rate of Non Vital Mature Anterior Teeth With Periapical Lesion Following Single Versus Two Visit Regenerative Treatment Protocol A Randomized Clinical Study
Brief Title: Success Rate of Single Versus Two Visit Regenerative Treatment Protocol in Non Vital Mature Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, lamiaa Mohamed Ragaei Lasheen, Assistant lecturer of endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faculty of dentistry 2018
Record Dates: First submitted 2018-10-14; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Pulp Necrosis; Periapical Lesion; Anterior Teeth
Keywords: Regeneration, mature teeth, regenerative procedures
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: The design of this randomized clinical trial is a parallel group two arms trial with 1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single visit pulp regeneration (Experimental): Regenerative endodontic procedure not involving placement of intracanal medicament will be done in single visit
  Interventions: Procedure: Single visit pulp regeneration
- Two visit pulp regeneration (Active Comparator): Regenerative endodontic procedure involving placing intracanal medicament will be done in two visit
  Interventions: Procedure: Two visit pulp regeneration

INTERVENTIONS:
Procedure: Single visit pulp regeneration — Access cavity, disinfection, preparing and injecting platelet rich plasma, and restoring the tooth all done in one visit.
  Arms: Single visit pulp regeneration
Procedure: Two visit pulp regeneration — first visit : access, disinfection and placing calcium hydroxide as intracanal medicament second visit: re opening of tooth, preparing and injecting platelet rich plasma and restoring the tooth.
  Arms: Two visit pulp regeneration

SUMMARY:
This study evaluates success rate of non vital mature anterior teeth with periapical lesion treated by regenerative endodontic protocol in single visit versus two visit technique.

Patients are randomized into two groups where treatment will be done either in one visit including access, disinfection, placing platelet rich plasma as scaffold and restoration or two visit protocol involving access, disinfection and placing calcium hydroxide as intracanal medicament in first visit followed by a second visit after 3 weeks involving reopening of the tooth, removing intracanal medicament and placing platelet rich plasma as scaffold then restoration. Success rate is defined as absence of subjective signs and symptoms along with healing of periapical lesion

DETAILED DESCRIPTION:
Title: Evaluation of Success Rate of Non Vital Mature Anterior Teeth with Periapical Lesion Following Single versus Two Visit Regenerative Treatment Protocol (A Randomized Clinical Trial) Regenerative endodontics can be defined as biologically based procedures designed to replace damaged structures, including dentin and root structures, as well as cells of the pulp-dentin complex.

The majority of endodontic patients are adults, thus the application of the tissue engineering concept to mature teeth could provide a biological treatment modality instead of the conventional one. In fact, several advantages were reported about regenerative procedures in well developed mature teeth. Reconstitution of the neurovascular system in root canals by pulp regeneration will provide pulp tissues with an immune system, which will function as the first line of defense against microbial challenge. Moreover, restoration of pulp dentine complex will protect the tooth during loading and mastication.

Different treatment protocols for pulp regeneration were reported in the literature regarding irrigation (type, concentration and time), intracanal medication, pulpal space barrier, incorporation and lack of scaffolds (blood clot, PRP,PRF, collagen) as well as recall visits.

Rationale for conducting the research and choice of comparators:

Multiple visits protocol has been the commonly used technique in regenerative endodontic procedures. It involves the placement of intracanal medicaments between visits (calcium hydroxide and triple antibiotic paste) which have many drawbacks such as difficulty in removal, tooth discoloration, weakening of the root and tooth loss.

Completing revascularization in one visit has many advantages. First, it reduces the chance of additional bacterial contamination of the space. Second, a single revascularization protocol may overcome the problem of poor patient compliance and reduce the number of appointments needed. Third, it can help to combat potential injury of the tooth and tooth discoloration Unfortunately, up till the moment it is not clear which protocol is the most effective. Thus randomized clinical trials are required to provide plausible answers to this question In the present research the recent single visit regenerative treatment for necrotic mature teeth will be compared to the conventionally used two visit one

ELIGIBILITY:
Inclusion Criteria:

* Single canal anterior tooth

  * Mature root
  * Non vital with radiographic evidence of periapical lesion
  * Periapical lesion of average size 2-5mm
  * Positive patient compliance for participation in the study.
  * Patients with good oral hygiene
  * Normal periodontal probing depth ≤ 3 mm

Exclusion Criteria:

* Compromised remaining tooth structure that need post and core build up
* Non restorable teeth
* Vital teeth
* Radiographic evidence of external or internal root resorption.
* Roots showing fracture or ankylosis
* Medically compromised patients
* Pregnant women
* Greater than grade I mobility or periodontal probing depth greater than 3mm
* Immature tooth
* Patients with pain, swelling or fistula tracts

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Post operative pain: NRS | 3, 6, 9 and 12 months
  absence of pain reported by the patient by numerical rate scale, the 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Change in swelling and/or sinus | 3,6,9,12 months
  The presence of swelling or sinus will be reported by a binary question yes/no
Periapical healing | 12 months
  The existing periapical lesion will be measured by mm by CBCT before intiation of treatment and after one year

SECONDARY OUTCOMES:
Antimicrobial effect | before and after complete disinfection either in the same visit or after 3 weeks from the second visit
  intracanal bacterial count by culture method
Sensitivity | 3, 6, 9 and 12 months
  Tooth giving respond to electrical pulp tester
Discoloration | 3, 6, 9 and 12 months
  Recording tooth shade before and after treatment

REFERENCES:
- [Derived] Lasheen LR, Gawdat SI, Lutfy RA. Success Rate of Single Versus Two-Visit Regenerative Treatment Protocol in Non-Vital Mature Anterior Teeth (A Preliminary Randomised Clinical Trial). Aust Endod J. 2025 Aug;51(2):308-316. doi: 10.1111/aej.12943. Epub 2025 Apr 11. PMID 40219648